CLINICAL TRIAL: NCT07172906
Title: "Nutrition Education by Nurses in Patients After Coronary Artery Bypass Grafting: Effect on Patients' Dietary Pattern, Adherence and Clinical Outcomes"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Mediterranean University (Other)
Collaborators: University General Hospital of Heraklion (Other)
Responsible Party: Principal Investigator, Konstantinos Giakoumidakis, Associate Professor, Department of Nursing, Hellenic Mediterranean University, Hellenic Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7736/20-02-2025
Record Dates: First submitted 2025-06-12; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Artery Bypass Grafting; Nutritional Education from nurses; Weight measurement; adherence to the Mediterranean diet
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Control Group) (Active Comparator): These are patients who will have their body measurements, weight, body fat and water percentage measured. They will also complete the questionnaires that will be included in the study, but they will not receive any nutritional education from the researcher.
  Interventions: Behavioral: Patients of Group A and B both are filling out the questionnaire "Mediterranean diet questionnaire (MEDAS)"; Behavioral: Patients of Group A and B both are filling out the "Mini Nutritional Asessment" questionnaire; Behavioral: Patients of Group A and B both are filling out "Nottingham Health Profile Scale" questionnaire; Behavioral: Patients of Group A and B both are filling out the "Cardiovascular Diet Questionnaire-2"; Other: Measurement of patient somatometric characteristics
- Intervention Group (Group B) (Active Comparator): These are patients who will have their body measurements, weight, body fat and water percentage measured. They will also complete the questionnaires that will be included in the study. These patients will receive nutritional education from the researcher, through an information sheet, phone calls and messages. The goal is to improve their measurements and their nutritional choices due to this education, compared to the patients in Group A.
  Interventions: Behavioral: Patients of Group A and B both are filling out the questionnaire "Mediterranean diet questionnaire (MEDAS)"; Behavioral: Patients of Group A and B both are filling out the "Mini Nutritional Asessment" questionnaire; Behavioral: Patients of Group A and B both are filling out "Nottingham Health Profile Scale" questionnaire; Behavioral: Patients of Group A and B both are filling out the "Cardiovascular Diet Questionnaire-2"; Other: Measurement of patient somatometric characteristics; Behavioral: Nutritional education and discussion with group B patients

INTERVENTIONS:
Behavioral: Patients of Group A and B both are filling out the questionnaire "Mediterranean diet questionnaire (MEDAS)" — This questionnaire will be completed by patients in both groups. The aim of this questionnaire is to assess the patients' dietary choices and how beneficial they are for their health, according to the Mediterranean diet model.
Behavioral: Patients of Group A and B both are filling out the "Mini Nutritional Asessment" questionnaire — This questionnaire will be completed by patients in both groups. The aim of this questionnaire is to assess the nutritional status of the patients, their level of nutrition and appetite for food, and the potential risk of malnutrition.
Behavioral: Patients of Group A and B both are filling out "Nottingham Health Profile Scale" questionnaire — This questionnaire will be completed by patients in both groups. The aim of this questionnaire is to assess the subjective discomfort of the individual with health problems as well as the extent to which these problems affect their normal activities.
Behavioral: Patients of Group A and B both are filling out the "Cardiovascular Diet Questionnaire-2" — This questionnaire will be completed by patients in both groups. The aim of this questionnaire is to assess the dietary choices of patients with cardiovascular diseases, such as the patients in this study.
Other: Measurement of patient somatometric characteristics — Measurement of body weight, Body Mass Index, Fat and Water Percentage, Chest, Waist and Hip Circumference of patients using a tape measure and electronic scale-lipometer. Also, measurement of bloodless blood pressure and fasting glucose.
Behavioral: Nutritional education and discussion with group B patients — Nutritional education using an information leaflet, e-mails and telephone calls to patients in group B only. Discussion regarding their dietary choices before surgery, identification of wrong habits and efforts to improve them afterwards. It will concern all the basic categories of healthy eating (preference for fruits, vegetables, proteins, healthy carbohydrates, reduction of saturated fat, salt and sugar and information about nutritional labels and how to choose foods according to them). The goal is for patients who will receive this education to improve their measurements in repeat meetings with the researcher, compared to those who will not be informed.
  Arms: Intervention Group (Group B)

SUMMARY:
The purpose of this study is the investigation of the effect of nurse-led nutritional education of post-CABG patients on their dietary pattern, on their adherence to it, but also on their quality of life and well-being.

DETAILED DESCRIPTION:
Introduction Cardiovascular disease is the leading cause of death worldwide, leading to approximately 18 million deaths annually. Coronary Artery Bypass Grafting (CABG) is the surgical treatment of coronary artery disease, which improves patients' symptoms and quality of life. However, successful postoperative recovery requires the adoption of a healthy lifestyle, including proper nutrition. Research shows that a diet high in unsaturated fat and low in saturated fat can improve the metabolic profile and cardiovascular function, reducing morbidity and potential complications. In addition, a balanced diet contributes to improving mental health and well-being, reducing anxiety and the occurrence of cognitive disorders such as postoperative delirium. Therefore, adherence to a healthy dietary pattern is crucial for the long-term management of the disease and the successful recovery of cardiac surgery patients.

Methodology A clinical study will be conducted with manipulation of independent variables and creation of a control group. Patients will be approached and randomly assigned to two groups: a) the control group (Group A), where patients will receive standard care based on the policy and protocols of the Tertiary Hospitals and b) the Intervention Group (Group B), where patients will receive nurse-led education through oral sessions, provision of an educational form and telephone calls at regular intervals.

The Greek versions of the Mediterranean Diet Screener (MEDAS), Mini Nutritional Assessment (MNA) and Nottingham Health Profile Scale questionnaires, while translation and weighting will be carried out in the Greek population for the Cardiovascular Diet Questionnaire 2 (CDQ-2). The above aims to assess patients' compliance with specific dietary habits, while the latter concerns primarily cardiac patients. Questionnaires will be completed by all patients at the initial meeting and after 1, 3 and 6 months. Training and objective measurements will be performed only on patients in the intervention group. The statistical analysis of the data will be done with the SPSS program (version 26) and using descriptive and inductive statistical analysis methods.

Expected Results The proposed thesis aims to highlight the importance of nurse-led nutrition education in the care of patients after CABG. Education, through a variety of formats such as oral sessions, printed materials, home visits and telephone calls, is expected to improve patient outcomes, reducing the chances of hospital readmissions and improving their quality of life. In addition, it is expected to strengthen their adherence to healthy eating habits, contributing to the secondary and tertiary prevention of cardiovascular disease, and to reduce morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients who underwent CABG and were discharged from the hospital in the previous 10 days
* Knowledge of reading and writing in Greek by the patients
* Provision of written informed consent by the patients for their participation in the study

Exclusion Criteria:

* History of psychiatric illness, recent history of alcohol and/or drug abuse, dementia or Alzheimer's disease
* Patients with comorbidities (diabetes mellitus, chronic renal failure, idiopathic inflammatory bowel disease, other gastrointestinal disorders, food allergies, etc.) that would justify the adoption of a special dietary pattern that is not identical to the proposed dietary pattern
* Patients with a preference for strict vegetarianism (vegan) and/or cultural-religious beliefs that do not allow the adoption of the proposed dietary pattern

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Improving dietary choices and habits of patients with Coronary Heart Disease who underwent coronary artery bypass surgery | 6 months from the first meeting
  Through nutritional education and discussion with the researcher, the goal is for patients to understand healthy eating choices, make better choices regarding their diet, and improve the outcome of surgery.

SECONDARY OUTCOMES:
Improvement in body weight (kg) of patients | Until 6 months from the first meeting with the researcher
  Through the nutritional education that patients will receive, they will be able to properly understand healthy dietary choices and improve their body weight (mainly overweight and obese patients will be able to reduce it to healthy limits). Their weight will be measured with an electronic scale.
Improving patients' Body Mass Index to healthy limits | 6 months from the first meeting
  Through the nutritional education that patients will receive, they will be able to properly understand healthy dietary choices and improve their Body Mass Index. Body mass index will be calculated using an electronic scale after body weight has been measured.
improvement of patients' body fat percentage (%) and body water percentage (%) | Until 6 months from the first meeting
  Due to improved dietary choices after training, patients will be able to improve their body fat and water percentage (especially overweight and obese patients). These parameters will be calculated with a special scale - lipometer, after measuring body weight and also calculating the patient's gender, age and height.
Improving patients' chest, waist and hip circumferences (cm) to healthy limits | Until 6 months from the first meeting
  In addition to improving the parameters of weight, fat, water and Body Mass Index, it is important to improve the measurements of the patients' chest, waist and hip circumferences to healthy limits (reduction in overweight and obese patients and increase in malnourished patients). This measurement will be done with a tape measure by the researcher.

IPD SHARING:
Plan to Share IPD: No
The data collected will be anonymous, used exclusively for the purposes of the research, and will be accessible only to the principal investigator. Participants will provide written consent, having been fully informed that the process is anonymous, their personal information and responses will be used exclusively for research purposes, and they can withdraw at any time. All data will be stored and will remain stored for as long as necessary until their analysis and then destroyed.